CLINICAL TRIAL: NCT00927121
Title: l Prospective Clinical Investigation on the Acoustic Stimulation With the "Coordinated Reset of Neural Subpopulations" in the Treatment of Chronic Tinnitus
Brief Title: Clinical Investigation on the Acoustic Stimulation in the Treatment of Chronic Tinnitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANM Adaptive Neuromodulation GmbH (Industry)
Responsible Party: Central Coordinating investigator: Prof. Dr. Dr. Peter Tass, Research Center Jülich, Institute for Neurosciences and Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/1525
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Tonal Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 : G_1 (Active Comparator): G_1: stimulation for 4 - 6 hours a day, 4 tones per sequence
  Interventions: Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset
- Group 2 :G_2 (Active Comparator): G_2: stimulation for 4 - 6 hours a day with 12-tone sequences
  Interventions: Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset
- Group3 : G_3 (Active Comparator): G_3: stimulation for 4 - 6 hours a day, 4 tones per sequence with a signal controlled by EEG measurement
  Interventions: Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset
- Group 4 : G_4 (Active Comparator): G_4: stimulation for 1 hour a day, 4 tones per sequence
  Interventions: Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset
- Group5 : G_5 (Placebo Comparator): G_5: stimulation with placebo-tone
  Interventions: Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset

INTERVENTIONS:
Device: Acoustic CR-Stimulator ANM//Technology: Acoustic coordinated reset — The CR-stimulation was originally developed by Prof. Dr. Dr. Peter Tass for deep brain stimulation (DBS). The CR-stimulation through high frequency short pulses causes a neuronal reorganization in the stimulated brain area establishing a normal neuronal activity.
  Based on intensive modeling studies, experimental proof of concept (POC) animal studies and a clinical POC, we proved that the pathologic activity can be recuperated to a desynchronized/healthy state with the acoustic CR-stimulation.
  The acoustic CR-stimulation signal will be generated by the ANM CR-Stimulator and transmitted to the ears through a speaker system

SUMMARY:
There are many treatments for chronic tinnitus that have been claimed, with varying degrees of statistical reliability. None of those treatments can eradicate the tinnitus completely. Some therapies can reduce the tinnitus symptoms (loudness, annoyance) up to 30%. Thus there is still a need of new treatments that can reduce considerably the tinnitus symptoms and improve the QOL of subjects.

Trial objectives:

* The aim of this trial is the improvement of the QOL (quality of live) by reducing the Tinnitus- Symptoms of the patient.
* To confirm the efficacy and safety of the coordinated reset technology.

These objectives will be assessed:

* By subjective and objective measurements of the Tinnitus symptoms, loudness and annoyance.

ELIGIBILITY:
Inclusion Criteria:

* Mentally healthy people
* Chronic tonal Tinnitus
* Older than 18 years
* Signature of the patient informed consent
* No participation in other tinnitus therapy during the clinical investigation

Exclusion Criteria:

* A necessity for hearing aid
* Auditory hallucination
* Symptomatic hearing disorders
* "Morbus Meniere",
* Tinnitus due to temporomandibular joint disorders
* Subjects who can't perceive therapeutic tones
* Brainstem diseases
* Psychiatric disorders
* Objective Tinnitus
* Insufficient treatment of general disorders, anemia, tumor, dialysis, hypertonus ect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Jülich // Institute for Neurosciences and Medicine - Research Center, Jülich, Germany

REFERENCES:
- [Result] Tass PA, Adamchic I, Freund HJ, von Stackelberg T, Hauptmann C. Counteracting tinnitus by acoustic coordinated reset neuromodulation. Restor Neurol Neurosci. 2012;30(2):137-59. doi: 10.3233/RNN-2012-110218. PMID 22414611
- [Derived] Adamchic I, Langguth B, Hauptmann C, Tass PA. Psychometric evaluation of visual analog scale for the assessment of chronic tinnitus. Am J Audiol. 2012 Dec;21(2):215-25. doi: 10.1044/1059-0889(2012/12-0010). Epub 2012 Jul 30. PMID 22846637
- See also: Counteracting tinnitus by acoustic coordinated reset neuromodulation. Tass PA, Adamchic I, Freund HJ, von Stackelberg T, Hauptmann C. — http://iospress.metapress.com/content/r771875822464323/?p=c8cb085557f04bd0b9c22d1d2e9d3eb6&pi=0